CLINICAL TRIAL: NCT03798353
Title: Pericardial Matrix With Mesenchymal Stem Cells for the Treatment of Patients With Infarcted Myocardial Tissue (The PERISCOPE Trial)
Brief Title: Pericardial Matrix With Mesenchymal Stem Cells for the Treatment of Patients With Infarcted Myocardial Tissue
Acronym: PERISCOPE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fundació Institut Germans Trias i Pujol (Other)
Collaborators: Germans Trias i Pujol Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICOR-2016-02; 2018-001964-49 (EudraCT Number)
Record Dates: First submitted 2018-12-21; First posted 2019-01-09 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-12

CONDITIONS: Myocardial Infarction
Keywords: Cardiac repair; Wharton jelly mesenchymal stem cells; Chronic myocardial infarction; Tissue engineering; Cell therapy; Clinical trial
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: - Experimental group: The patient will undergo surgery by sternotomy to perform the surgical revascularization of the arteries candidates for revascularization.
  In addition, the matrix-cell construct will be placed on the ischemic area of the non-candidate revascularization area and will be fixed using surgical glue.
  - Control group: The patient will undergo surgery by sternotomy to perform the surgical revascularization of the arteries candidates for revascularization. No additional procedure will be performed.
Who Masked: Participant, Investigator
Masking Description: The randomization will be known exclusively by the cardiac surgery team and the study coordinator, and it will be blind to the patient and to the rest of the investigators team: clinical cardiologist who performs the follow-up, team that performs image tests, core lab that evaluates the imaging tests and the equipment that statistically analyzes the data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The patient will undergo surgery by sternotomy to perform the surgical revascularization of the arteries candidates for revascularization.
  In addition, the matrix-cell (PeriCord) construct will be placed on the ischemic area of the non-candidate revascularization area and will be fixed using surgical glue.
  PeriCord: Expanded and cryopreserved allogeneic umbilical cord Wharton´s jelly-derived adult mesenchymal stem cells colonized on human pericardial matrix .
  Interventions: Combination Product: PeriCord: Expanded and cryopreserved allogeneic umbilical cord Wharton´s jelly-derived adult mesenchymal stem cells colonized on human pericardial matrix.
- Control group (Active Comparator): The patient will undergo surgery by sternotomy to perform the surgical revascularization of the arteries candidates for revascularization. No additional procedure will be performed.
  Interventions: Procedure: Surgery by sternotomy

INTERVENTIONS:
Combination Product: PeriCord: Expanded and cryopreserved allogeneic umbilical cord Wharton´s jelly-derived adult mesenchymal stem cells colonized on human pericardial matrix. — A matrix-cell construct (PeriCord) will be placed on the ischemic area of the non-candidate revascularization area during a surgery by sternotomy to perform the surgical revascularization of the arteries candidates for revascularization.
  Arms: Experimental group
Procedure: Surgery by sternotomy — The patient will undergo surgery by sternotomy to perform the surgical revascularization of the arteries candidates for revascularization. No additional procedure will be performed only the by-pass.
  Arms: Control group

SUMMARY:
Myocardial infarction causes necrosis of myocardial cells and reduces cardiac function. Today, there are treatments such as primary angioplasty and thrombolysis that are effective in limiting cell death after acute myocardial infarction. However, the post-infarct scar often conditions a global ventricular remodeling that can evolve clinically towards heart failure and in more advanced stages the only therapy that completely restores cardiac function is heart transplantation.

Mesenchymal stem cells are multipotent cells found from embryonic mesoderm and found in all tissues. In the field of cardiac regeneration, studies have shown a certain degree of benefit when treated with MSCs from different origins. Our approach is based on a decellularized matrix that carries the cells directly over myocardial infarction.

DETAILED DESCRIPTION:
Myocardial infarction causes necrosis of myocardial cells and reduces cardiac function. Today there are treatments such as primary angioplasty and thrombolysis that are effective in limiting cell death after acute myocardial infarction. However, the post-infarct scar often conditions a global ventricular remodeling that can evolve clinically towards heart failure and, in more advanced stages, the only therapy that completely restores cardiac function is heart transplantation.

Experimental studies are evaluating new therapeutic approaches based on tissue engineering for myocardial regeneration. Cardiac tissue engineering attempts to create functional tissue constructs that can restore the structure and function of damaged myocardium.

Mesenchymal stem cells (MSCs) are multipotent cells that develop from embryonic mesoderm and are found in all structural tissues of the body.

In the field of cardiac regeneration, studies have shown a certain degree of benefit when treated with MSCs from different origins. The investigators approach is based on a decellularized matrix that carries the cells directly over myocardial infarction.

Among the different types of MSC currently available, the investigators propose the use of those derived from the connective tissue surrounding the great vessels (2 arteries and one vein) of the umbilical cord called Wharton's gelatin (MSC, WJ) whose immunomodulatory properties are described extensively in the literature. These MSC, WJ cells have a PEI approved by the Spanish Agency for Medicines and Healthcare Products (AEMPS) (PEI 16-017) that guarantees an optimal manufacturing process for a clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Myocardial infarction of ≥50% of transmurally due to MR
* Candidate for coronary by-pass through that or another territory
* Age ≥18 years
* Signature of informed consent
* Wave Q present in the ECG
* Followed by the cardiology service of Germans Trial i Pujol hospital

Exclusion Criteria:

* Severe valvular disease with indication of surgical repair
* Candidate for ventricular remodeling
* Contraindication for MR (creatinine clearance less than 30 ml / min / 1.73m2, metallic implant carriers, claustrophobia)
* Extracardiac disease with estimated life expectancy less than 1 year
* Neoplastic disease detected in the last five years or without complete remission
* Severe renal or hepatic insufficiency
* Abnormal laboratory values, not explainable at the time of inclusion, and that at the discretion of the investigator contraindicate the patient's participation in the study
* Patients with a previous cardiac intervention
* Women who are pregnant or breast-feeding.
* Women of childbearing age who are heterosexually active and who do not use an effective contraceptive method from 14 days before the inclusion in the study and at least up to 12 weeks after the end of the study.
* Simultaneous participation in another clinical trial or treatment with another product in investigational phase in the 30 days prior to inclusion in the study.
* Negation of the patient to be followed by a period that exceeds the clinical trial itself (long-term follow-up in the second and third year).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2022-10-06 (Actual)

PRIMARY OUTCOMES:
Rate of death or rehospitalization due to any cause and / or adverse reactions related to the procedure / product under investigation. | at 12 months of follow-up
  Safety measured with a combined endpoint of serious clinical events (death or rehospitalization due to any cause) and serious adverse reactions related to the investigational treatment.

SECONDARY OUTCOMES:
Rate of death or rehospitalization due to any cause and / or adverse reactions related to the procedure / product under investigation. | At 1 week, 3 and 6 months
  Safety measured with a combined endpoint of serious clinical events (death or rehospitalization due to any cause) and serious adverse reactions related to the investigational treatment
Death rate or rehospitalization due to cardiovascular causes | At 1 week, 3 , 6and 12 months
  Death rate or rehospitalization due to cardiovascular causes at week, 3, 6 and 12 months.
Rate of relevant arrhythmias in Holter of 24 hours | At 1 week, 3 and 12 months
  Rate of relevant arrhythmias in Holter of 24 hours a week, 3 and 12 months.
Relevant changes in N-terminal B-type natriuretic peptide (NT-proBNP) and High sensitivity troponin I (hsTnI) levels | At 1 week, 3 and 12 months
  Relevant changes in NT-proBNP and hsTnI levels at week, 3 and 12 months.
Changes in the necrotic myocardial mass ratio | At 3 and 12 months
  Changes in the necrotic myocardial mass ratio due to gadolinium retention at 3 and 12 months.
Changes of regional contractility | At 3 and 12 months
  change of regional contractility by nuclear magnetic resonance (NMR) at 3 and 12 months.
Changes in ejection fraction of the left ventricle | At 3 and 12 months
  Changes in ejection fraction of the left at 3 and 12 months
changes in left and right ventricular geometric remodeling | At 3 and 12 months
  changes in left and right ventricular geometric remodeling at 3 and 12 months
Changes in the score on the quality of life test Short Form 36 Healthy Survey (SF-36). | At 3 and 12 months
  Changes in the score on the quality of life test SF-36 will be used at 3 and 12 months. The mínimum value is 0 and the máximum value is 100. Higher scores mean a better outcome.
Changes in the score on the quality of life Kansas City Cardiomyopathy Questionnaire (KCCQ) test in cases of participants with heart failure will be used. | At 3 and 12 months
  Changes in the score on the quality of life test KCCQ in cases of participants with heart failure will be used at 3 and 12 months. The test is composed of 23 items. The options for the answers are Likert scales of 1 to 5, 6 or 7 points and the score of each of its dimensions has a theoretical range from 0 to 100, 100 being the best outcome.

OTHER OUTCOMES:
monocyte populations and cytokines and chemokines levels | At screening, day 3 and day 5
  changes in the monocyte populations and cytokines and chemokines levels between the two groups in order to analyze if the PeriCord could improve these variables

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Bayes-Genís, MD, PhD,FESC, Principal Investigator — Institut del Cor, HUGTiP, IGTP
Locations (1):
- Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona, Spain